CLINICAL TRIAL: NCT01328717
Title: Clinical Trial Protocol for Contour Link System With Contour Sensor
Brief Title: Performance of an Investigational Blood Glucose Monitoring System in a Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R&D-2010-2011.09
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the System (Experimental): Subjects with diabetes used Contour Link Investigational Blood Glucose Monitoring System
  Interventions: Device: Contour Link Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Contour Link Investigational Blood Glucose Monitoring System — Subjects with diabetes and study staff each performed Blood Glucose tests from the subject's capillary blood obtained from fingerstick using the Contour Link investigational meter.

SUMMARY:
Subjects with diabetes and study staff used an investigational blood glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and above
* Diagnosed as having type 1 or type 2 diabetes
* Currently self-testing blood glucose at home for at least three months
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Gestational Diabetes
* Hemophilia or any other bleeding disorder
* Employee of competitive medical device company

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the System: Subjects with diabetes and study staff used an investigational blood glucose monitoring system. As a result of one subject's low blood sugar (and thus rapidly changing glucose values) during the study, 77 subjects completed the study.
Period: Overall Study
Arm/Group | Intended Users of the System
Started | 78
Completed | 77
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 77
Age, Customized [Mean (Full Range); unit: years] | 55 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Percent of Fingerstick Blood Glucose (BG) Results Within +/-20%(>=75 mg/dL) and Within +/- 15mg/dL (<75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes and study staff tested subject fingerstick blood using an investigational blood glucose meter (BGM). BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 20% (for reference BG results >=75mg/dL) and within +/- 15mg/dL(for reference BG results <75mg/dL) of the reference method results.
Time Frame: 1 hour
Population: As a result of one subject's low blood sugar (and thus rapidly changing glucose values) during the study, one subject did not complete the study. The remaining 77 subjects tested 2 test strip lots on the system. 2x77(154) test results were available.
Measure: Number; unit: Percentage of BG test results
Units Other Than Participants: Blood Glucose Test Results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 77
Number analyzed (Blood Glucose Test Results) | 154
Percentage of BG test results | 95.5

2. Secondary Outcome: Number of Subjects Rated as<=3 Performing Basic Meter Tasks (Labeling Evaluation)
Description: Subjects read User Guide(UG)to learn to use the system and performed meter tasks. Study staff observed, then rated subjects' success (1 to 4) at performing tasks. Scale: 1.Performed tasks correctly without assistance. 2.Performed tasks correctly, but was directed to a specific part of the UG by the study staff as in a Customer Service call. 3.Performed tasks correctly, but required additional review/assistance similar to review of a specific function during a Customer Service call. 4.Subject incorrectly performed part of the testing regimen and was unaware of the error.
Time Frame: 1 hour
Population: Per protocol
Measure: Number; unit: Number of Participants
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 77
Number of Participants
  Turn meter on and off | 77
  Set meter time and date | 77
  Perform fingerstick blood test | 77
  Perform control test | 77

ADVERSE EVENTS:
Arm/Group | Intended Users of the System
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 2/78
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the System (N=78)
hypoglycemia (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes